CLINICAL TRIAL: NCT05991908
Title: Multiple-center Randomized Study to Compare Fludarabine and Busulfan Versus Fludarabine, Busulfan and Melphalan in Adult Patients With Acute Myeloid Leukemia (AML) and Myelodysplasia Syndrome (MDS)
Brief Title: Randomized Study of Conditioning of Fludarabine Combined With Single or Dual Alkylating Agents in Myeloid Malignancies
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBF-FB4
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: conditioning regimen, melphalan, busulfan, fludarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine; Busulfan; Melphalan

STUDY DESIGN:
Intervention Model Description: study group with fludarabine, busulfan and melphalan regimen versus control group with fludarabine and busulfan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flu-Bu2-Mel140 (Experimental): Patients receive fludarabine, busulfan and melphalan as conditioning regimen
  Interventions: Drug: Fludarabine, busulfan and melphalan
- Flu-Bu4 (Active Comparator): Patients receive fludarabine and busulfan as conditioning regimen
  Interventions: Drug: Fludarabine and Busulfan

INTERVENTIONS:
Drug: Fludarabine, busulfan and melphalan — FLudarabine 150mg/m2 + Busulfan 6.4mg.kg + Mel 140mg/m2
  Arms: Flu-Bu2-Mel140
Drug: Fludarabine and Busulfan — FLudarabine 150mg/m2 + Busulfan 12.8mg.kg
  Arms: Flu-Bu4

SUMMARY:
Fludarabine and busulfan becomes standard conditioning regimen for adult patients with acute myeloid leukemia (AML) or myelodysplasia syndrome (MDS). The overall relapse rate is 15~20%. More recently, the investigators demonstrated that conditioning regimen with dual alkylating agents consistent of fludarabine, busulfan and melphalan achieved a low incidence of relapse (<10%). This multiple-center randomize study is aim to compare the transplantation outcome in adult patients with AML/MDS undergoing allo-HSCT with conditioning regimen of Flu-Bu4 vs. FLu-Bu-Mel.

DETAILED DESCRIPTION:
Fludarabine and busulfan was considered as myeloablative but reduced toxicity regimen and became as the mainstay of conditioning regimen for adult patients with acute myeloid leukemia (AML) or myelodysplasia syndrome (MDS). The disease relapse remained as major cause of treatment failure. In general, the cumulated incidence of relapse (CIR) is about 15~20% dependent on the risk of patients undergoing allogeneic stem cell transplantation (allo-HSCT). Conditioning regimen with dual alkylating agents such as fludarabine, busulfan and thiotepa (TBF) showed decreased risk of relapse in myeloid malignancies. More recently, the investigators demonstrated that conditioning regimen with dual alkylating agents consistent of fludarabine, busulfan and melphalan could achieve a low incidence of relapse (2 year CIR <10%). In this multiple-center randomize study, the aim is to compare the transplantation outcome in adult patients with AML/MDS undergoing allo-HSCT with conditioning regimen of Flu-Bu vs. Flu-Bu-Mel.

ELIGIBILITY:
Inclusion Criteria:

* acute myeloid leukemia (acute promyelocytic leukemia excluded) in 1st complete remission
* myelodysplasia syndrome with bone marrow blast >5% and remaining less than 20% at transplantation
* patients with HLA matched sibling donor, 9-10 matched unrelated donor or haplo-identical related donors
* inform consent provided

Exclusion Criteria:

* AML patients with active CNS or extramedullary diseases
* patients with active viral, bacterial or fungal infection
* patients with hepatitis B virus >1X103 copy/ml
* patients with abnormal liver function, renal function, respiratory or cardiac dysfunction
* patients with uncontrolled mental disorders
* patients with HIV

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 222 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 2 year
  event defined as relapse and death of any causes

SECONDARY OUTCOMES:
overall survival | 2 year
  event defined as death of any causes
incidence of relapse | 2 year
  event defined as disease relapse (bone marrow or extra medullary)
non relapse mortality | day 100
  event defined as death without disease relapse
non relapse mortality | 2 year
  event defined as death without disease relapse

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, Principal Investigator — Go Broad Health Center, Zhaxin Hospital
Locations (9):
- China (9):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Zhongshan Hospital, Xianmen University, Xiamen, Fujian
  - 923th Hospital PLA, Nanning, Guangxi
  - First Affiliated Hospital of Nanjin Medical Unviersity, Nanjin, Jiangsu
  - First Affiliatied Hospital of Soochow University, Suzhou, Jiangsu
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai No10 Hospital, Shanghai, Shanghai Municipality
  - 920th Hospital PLA, Kunming
  - Shanghai No 6 Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No